CLINICAL TRIAL: NCT03231072
Title: Effects of the Pleural Effusion Drainage in Mechanically Ventilated Patients Monitored by Electrical Impedance Tomography and End-Expiratory Lung Volume
Brief Title: Pleural Effusion Drainage in Mechanically Ventilated Patients Monitored by EIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Czech Technical University in Prague (Other)
Collaborators: Military University Hospital, Prague (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Ventilation-EIT-PE
Record Dates: First submitted 2017-07-18; First posted 2017-07-27 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Pleural Effusion; Drainage; Electric Impedance Tomography
Keywords: mechanical ventilation; pleural effusion; EIT
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Electrical Impedance Tomography record (Experimental): Electrical Impedance Tomography monitoring of the pleural effusion evacuation.
  Interventions: Device: Electrical Impedance Tomography record

INTERVENTIONS:
Device: Electrical Impedance Tomography record — Monitoring of pleural effusion evacuation by means of EIT

SUMMARY:
Evacuation of pleural effusion (PE) represents a disputable therapy in mechanically ventilated patients. Patients on mechanical ventilation indicated by the physician to pleural fluid evacuation will be monitored throughout the procedure by electrical impedance tomography (EIT) and concurrently end-expiratory lung volume (EELV) will be measured in order to describe impact of PE evacuation on aeration and ventilation of the lungs.

DETAILED DESCRIPTION:
Critically ill patients treated in intensive care units have a disorder of distribution and volume of body fluids due to principal illness and some therapeutic interventions. One of its manifestations is pleural effusion (PE) formation.

Patients on mechanical ventilation indicated by treating physician to pleural fluid evacuation will be monitored throughout the procedure by electrical impedance tomography (EIT) and concurrently end-expiratory lung volume (EELV) will be measured. The purpose of the study is to better understand impact of PE evacuation on aeration and ventilation of the lungs.

ELIGIBILITY:
Inclusion Criteria:

* mechanical ventilation, presence of pleural effusion, decision of the treating physician to drain it

Exclusion Criteria:

* impossibility to apply EIT belt or to find suitable save point for drainage when the EIT belt is attached
* standard EIT exclusion criteria according to the device manufacturer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Change of the thorax electrical impedance following pleural effusion drainage in mechanically ventilated patients | 4 hours
  Comparison of EIT results with end-expiratory lung volume measurement during drainage of pleural effusion

SECONDARY OUTCOMES:
Change of the distribution of ventilation following pleural effusion drainage in mechanically ventilated patients | 4 hours
  Change of distribution of ventilation over EIT regions of interest (ROIs)

CONTACTS AND LOCATIONS:
Overall Officials: Karel Roubik, Prof., PhD., Principal Investigator — Czech Technical University in Prague
Locations (1):
- The Military University Hospital, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Razazi K, Thille AW, Carteaux G, Beji O, Brun-Buisson C, Brochard L, Mekontso Dessap A. Effects of pleural effusion drainage on oxygenation, respiratory mechanics, and hemodynamics in mechanically ventilated patients. Ann Am Thorac Soc. 2014 Sep;11(7):1018-24. doi: 10.1513/AnnalsATS.201404-152OC. PMID 25079591
- [Background] Mattison LE, Coppage L, Alderman DF, Herlong JO, Sahn SA. Pleural effusions in the medical ICU: prevalence, causes, and clinical implications. Chest. 1997 Apr;111(4):1018-23. doi: 10.1378/chest.111.4.1018. PMID 9106583
- [Background] Goligher EC, Leis JA, Fowler RA, Pinto R, Adhikari NK, Ferguson ND. Utility and safety of draining pleural effusions in mechanically ventilated patients: a systematic review and meta-analysis. Crit Care. 2011;15(1):R46. doi: 10.1186/cc10009. Epub 2011 Feb 2. PMID 21288334
- [Background] Alves SH, Amato MB, Terra RM, Vargas FS, Caruso P. Lung reaeration and reventilation after aspiration of pleural effusions. A study using electrical impedance tomography. Ann Am Thorac Soc. 2014 Feb;11(2):186-91. doi: 10.1513/AnnalsATS.201306-142OC. PMID 24308560